CLINICAL TRIAL: NCT07256522
Title: Comparative Evaluation of Finger Splint, Paraffin, and Peloidotherapy Interventions in the Management of Trigger Finger. A Prospective, Randomized, Controlled Study
Brief Title: Comparative Evaluation of Finger Splint, Paraffin, and Peloidotherapy Interventions in the Management of Trigger Finger
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Konya Beyhekim Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Ramazan Yılmaz, MD, Associate Prof (MD), Konya Beyhekim Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KonyaBeyhekimTRH2025/5634
Record Dates: First submitted 2025-11-20; First posted 2025-12-01 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Trigger Finger; Splint Therapy; Paraffin Bath; Peloidotherapy; Efficacy and Safety; Randomised Clinical Trial
Keywords: trigger finger; splint therapy; paraffin bath; peloidotherapy; Randomised Controlled Study
MeSH Terms: conditions — Trigger Finger Disorder

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: single blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Finger orthosis (Experimental): The group receiving the finger joint-blocking orthosis
  Interventions: Device: Finger orthosis
- Paraffin bath (Experimental): The group receiving paraffin bath therapy
  Interventions: Other: Paraffin bath
- Peloidotherapy (Experimental): The group receiving peloidotherapy
  Interventions: Other: Peloidotherapy

INTERVENTIONS:
Device: Finger orthosis — Joint-blocking finger orthosis plus home-based exercise therapy
  Arms: Finger orthosis
Other: Paraffin bath — Paraffin bath plus home-based exercise therapy
  Arms: Paraffin bath
Other: Peloidotherapy — Peloidotherapy plus home-based exercise therapy
  Arms: Peloidotherapy

SUMMARY:
Patients aged 18-75 years who present with trigger finger to a tertiary rehabilitation hospital and agree to participate will be included in the study. Participants will be randomly allocated into three groups using block randomization. The first group will use a static finger splint that blocks the proximal interphalangeal joint for 6 weeks, along with a home exercise program. The second group will receive paraffin bath therapy, and the third group will receive peloidotherapy, both in combination with home exercises.

All patients will receive education about the disease and activity modification. The finger joint-restricting splint and exercises will be applied for 6 weeks. Evaluations will be conducted at baseline, at the end of the 3rd week, and at the end of the 6th week by a blinded assessor. No analgesic or anti-inflammatory medication will be permitted during the study, and patients will be instructed to avoid using analgesics within 24 hours prior to each assessment.

DETAILED DESCRIPTION:
Patients aged between 18 and 75 years who were diagnosed with trigger finger and agreed to participate in the study will be included. A total of 60 patients who have applied to the Physical Medicine and Rehabilitation outpatient clinics of the University of Health Sciences Beyhekim Training and Research Hospital will be enrolled. According to the inclusion and exclusion criteria, eligible and willing participants will be randomly assigned to three groups using block randomization.

The first group will be instructed to use a static finger splint that blocks the proximal interphalangeal joint for 6 weeks and will also follow a home exercise program. The second group will receive paraffin bath therapy for 20 minutes per day, 15 sessions over 3 weeks, together with a home exercise program. The third group will receive peloidotherapy at 45°C for 20 minutes per day, consisting of 15 sessions over 3 weeks, in conjunction with a home exercise program.

A static finger splint that restricts the proximal interphalangeal joint and maintains it in extension will be provided to the patients. They will be instructed to wear the splint continuously during both day and night, removing it only for hygiene or essential needs. The splint will be worn for 6 weeks until the completion of the study, and the daily duration of splint use will be recorded for each patient.

The home exercise program will include finger passive and active range of motion exercises (passive fist-making and active range of motion without triggering), tendon gliding, self-administered gentle A1 pulley stretching, and gentle deep circular massage. The exercises will be demonstrated to each patient in practice by a physician or physiotherapist and taught using printed visual materials. Patients will be specifically instructed, encouraged, and monitored to ensure exercise adherence. Those with an adherence rate below 70-75% will be excluded from the study.

All patients will receive education about the disease and will be advised on activity modification. Evaluations will be performed before treatment, at the end of the 3rd week, and at the end of the 6th week. A blinded assessor will conduct detailed examinations and evaluate the groups in terms of the study's primary and secondary outcome measures.

Patients' baseline sociodemographic and clinical data will be recorded, and a detailed physical examination will be performed. Pain intensity, trigger frequency, severity, and functional impact will be evaluated using a 0-10 Visual Analog Scale (VAS). Clinical staging of the trigger finger will be determined according to Green's classification (Grades 1-4). Patient compliance with orthotic use and exercise will be documented. Ultrasound assessments, including tendons thickness, A1 pulley thickness, and the presence of effusion (semiquantitative) will be performed by a blinded researcher with over five years of experience in musculoskeletal ultrasonography. In addition, patients' satisfaction levels will be evaluated and recorded using the Patient Global Improvement Scale. Any potential treatment-related undesirable effects effects will also be documented.

No analgesic or anti-inflammatory medication will be prescribed during the treatment period. Additionally, patients will be informed not to take any analgesic medication within 24 hours before the assessments.

ELIGIBILITY:
Inclusion Criteria:

* Being between 18 and 75 years of age and willing to participate in the study
* Having a diagnosis of idiopathic single trigger finger, Grade 2-3

Exclusion Criteria:

* Patients with triggering in more than one finger
* Patients with triggering at the A3 pulley or with Grade 1 or Grade 4 trigger finger
* Patients with thumb (pollex) trigger finger
* Patients who have undergone any injection or interventional procedure (release surgery) for trigger finger within the past 6 months
* Patients who have received physical therapy for the hand within the past 6 months
* Patients currently using corticosteroids or nonsteroidal anti-inflammatory drugs (NSAIDs)
* Patients with inflammatory or autoimmune rheumatologic diseases such as rheumatoid arthritis, systemic lupus erythematosus, gout, or psoriatic arthritis
* Patients with other musculoskeletal disorders (e.g., carpal tunnel syndrome, de Quervain's tenosynovitis, symptomatic hand osteoarthritis, or Dupuytren's contracture) or neurological diseases (e.g., stroke-related hemiparesis, spinal cord injury, brachial plexus injury, multiple sclerosis, or Parkinsonism) affecting the same hand
* Patients with musculoskeletal disorders causing pain and/or limitation in the proximal upper extremity on the affected side (e.g., periarthritis, lateral epicondylitis, mononeuropathy, or radiculopathy)
* Patients with significant metabolic diseases (e.g., hypothyroidism, Cushing's syndrome, or uncontrolled diabetes)
* Patients with any condition that may interfere with treatment, such as open wounds, rashes, local infections, or active malignant disease of the hand
* Patients with a history of hand trauma (chronic or repetitive)
* Patients unwilling to complete the self-assessment questionnaires either independently or with assistance
* Pregnant women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-11-03 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
VAS pain | Baseline, week 3 and week 6
  VAS pain: 0 no pain; 10 unbearable/max. pain.
Green's classification (Grades 1-4) | Baseline, week 2 and week 6
  Trigger finger classified according to Green's classification (Grades 1-4) Grade 1 - Pretriggering: Pain in the palm and tenderness over the A1 pulley, with a history of triggering not demonstrable on examination.
  Grade 2 - Active Triggering: Triggering is clinically evident, but the patient can actively extend the finger.
  Grade 3 - Passive Triggering:
  3a: Locking is present and requires passive extension.
  3b: Locking is present, and the patient cannot actively flex the finger.
  Grade 4 - Contracture: The finger is completely locked with a fixed flexion contracture at the PIP joint.
Michigan Hand Outcomes Questionnaire (MHQ) | Baseline, week 2 and week 6
  The Michigan Hand Outcomes Questionnaire (MHQ) is a comprehensive self-reported questionnaire developed to evaluate hand function, pain, and patient satisfaction. It is used to assess the functional status of individuals with upper extremity disorders and consists of six subscales: Overall Hand Function, Activities of Daily Living, Work Performance, Pain, Aesthetics, and Satisfaction. The Turkish version of the MHQ has undergone linguistic and cultural adaptation processes, and its validity and reliability have been established. Studies have demonstrated that the Turkish MHQ has high internal consistency and test-retest reliability, supporting its use in both clinical practice and research for assessing hand and wrist problems. The MHQ is scored on a scale ranging from 1 to 100. Except for the pain subscale, higher scores indicate better hand function and satisfaction, whereas higher pain scores represent greater pain intensity. The overall hand health status is determined by cal

SECONDARY OUTCOMES:
Patient Global Impression of Change | Week 2 and week 6
  Patient Global Impression of Change (Improvement):
  1: Very much improved 2: Much improved 3: Minimally improved 4: No change 5: Minimally worse 6: Much worse 7: Very much worse
Ultrasonographic evaluation of the trigger finger | Baseline, week 2 and week 6
  Ultrasonographic evaluation of the trigger finger will be performed using a LA2-14A transducer. The hand and forearm will be positioned with the palmar surface facing upward (full supination) and the wrist maintained in a neutral position. The ultrasound examination will begin in the longitudinal plane and then proceed to the transverse plane. The MCP joint, flexor tendons, and volar will be identified. At the level of the MCP joint, the transducer will be rotated to obtain a transverse image along the long axis of the flexor digitorum tendons. The thin layer located between the hyperechoic A1 pulley and the hyperechoic surface of the flexor digitorum tendons will represent the synovial fluid space, appearing as a hypoechoic band on ultrasonography. The thickness of the A1 pulley will be defined as the distance between its superior and inferior margins, including the hyperechoic region. The maximum thickness of the A1 pulley above the MCP joint will be measured and recorded.
Ultrasonographic evaluation of the trigger finger | Baseline, week 2 and week 6
  The cross-sectional areas (CSAs) of the flexor digitorum tendons will also be measured using a similar approach as described above. At the level of the MCP joint, the maximum CSAs of the flexor digitorum tendons will be manually traced in the transverse view along the outer hyperechoic contour. The average of three measurements will be calculated and recorded. Similar measurements will be performed on the corresponding finger of the contralateral healthy hand and recorded for comparison.

CONTACTS AND LOCATIONS:
Overall Officials: Ramazan Yilmaz, Assoc Prof, Principal Investigator — Konya Beyhekim Training and Research Hospital
Locations (1):
- Konya Beyhekim Training and Research Hospital, Konya, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No